CLINICAL TRIAL: NCT02040831
Title: A Phase I Study of the Safety and Immunogenicity of a Single Dose of the Recombinant Live-Attenuated Respiratory Syncytial Virus Vaccine RSV LID ΔM2-2, Lot RSV#007A, Delivered as Nose Drops to RSV-Seronegative Infants and Children 6 to 24 Months of Age
Brief Title: Safety and Immune Response to a Live-Attenuated Respiratory Syncytial Virus (RSV) Vaccine in RSV-Seronegative Infants and Children
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CIR 291
Record Dates: First submitted 2014-01-17; First posted 2014-01-20 (Estimated); Last update posted 2016-12-21 (Estimated); Status verified 2016-12

CONDITIONS: Respiratory Syncytial Virus Infections
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RSV LID ΔM2-2 Vaccine (Experimental): Participants will receive one dose of the RSV LID ΔM2-2 vaccine at study entry, delivered as nose drops.
  Interventions: Biological: RSV LID ΔM2-2 Vaccine
- Placebo Vaccine (Placebo Comparator): Participants will receive one dose of placebo at study entry, delivered as nose drops.
  Interventions: Biological: Placebo Vaccine

INTERVENTIONS:
Biological: RSV LID ΔM2-2 Vaccine — 10^5.0 plaque forming units (PFU); 0.5 mL dose delivered as nose drops (approximately 0.25 mL per nostril)
  Arms: RSV LID ΔM2-2 Vaccine
Biological: Placebo Vaccine — 0.5 mL dose delivered as nose drops (approximately 0.25 mL per nostril)
  Arms: Placebo Vaccine

SUMMARY:
Respiratory syncytial virus (RSV) is a common cause of illness in infants and children around the world. This study will evaluate the safety and immune response to an RSV vaccine in RSV-seronegative infants and children.

This study is a companion study to IMPAACT 2000.

DETAILED DESCRIPTION:
RSV is the most common viral cause of serious acute lower respiratory illness (LRI) in infants and children under 5 years of age in the world. RSV illness can range from mild upper respiratory tract illness (URI) to severe LRI, including bronchiolitis and pneumonia. Severe RSV disease in infancy may also predispose children to develop reactive airway disease during childhood. The purpose of this study is to evaluate the safety and immunogenicity of an RSV vaccine (RSV LID ΔM2-2) in RSV-seronegative infants and children at least 6 months and through 24 months of age.

To determine study eligibility, the screening process will include a blood collection. At study entry, eligible participants will be randomly assigned to receive one dose of either the RSV vaccine or placebo, which will be delivered as nose drops. Participants will also undergo a review of medical history, clinical assessment, and a nasal wash. They will then receive their assigned vaccine and will remain under observation for monitoring for 30 minutes after receiving the vaccine. Additional study visits will occur at Days 3, 5, 7, 10, 12, 14, 17, 19, 21, 28, and 56. These visits will include clinical assessments and nasal washes; on Day 56, a blood collection will also occur. On days where no study visit is scheduled (through Day 27), participants' parents or guardians will report participants' temperatures and signs of illness to researchers by e-mail or phone.

In October following vaccination, participants may have a pre-RSV season blood collection visit. During RSV season, November through March following vaccination, researchers will contact participants' parents or guardians on a weekly basis for follow-up monitoring. During this time frame, participants seen by a medical provider for fever, respiratory illness, or otitis media will have a study visit, which will include a nasal wash and clinical assessment. In April following vaccination, participants will undergo a final blood collection.

ELIGIBILITY:
Inclusion Criteria:

* Participant is at least 6 months but less than 25 months of age at the time of inoculation
* Parent or guardian who demonstrates their understanding of the study, signs the informed consent, and agrees to vaccine administration following detailed explanation of the study
* Seronegative for RSV antibody, defined as a serum RSV neutralizing antibody titer less than 1:40 as determined within 42 days prior to inoculation
* Participant's history has been reviewed and participant has undergone a physical examination indicating that s/he is in good health. Permitted concomitant medications include nutritional supplements, medications for gastroesophageal reflux, eye drops, and topical medications, including topical steroids, topical antibiotics, and topical antifungal agents.
* Participant has received routine immunizations appropriate for age, administered:

  1. at least 2 weeks prior to study vaccine inoculation (inactivated and subunit vaccines and rotavirus vaccine) OR
  2. at least 4 weeks prior to study vaccine inoculation (all other live vaccines)
* Participant is expected to be available for the duration of the study

Exclusion Criteria:

* Known or suspected impairment of immunological functions, including maternal history of positive HIV test
* Receipt of immunosuppressive therapy including systemic corticosteroids within the past 30 days. NOTE: Topical steroids, topical antibiotics, and topical antifungal medications are acceptable.
* Bone marrow/solid organ transplant recipient
* Major congenital malformations, including congenital cleft palate, cytogenetic abnormalities, or serious chronic disorders
* Previous immunization with an RSV vaccine
* Previous serious vaccine-associated AE or any anaphylactic reaction
* Known hypersensitivity to any vaccine component
* Lung or heart disease, including any wheezing event or reactive airway disease. NOTE: Participants with clinically insignificant cardiac abnormalities requiring no treatment may be enrolled. Participants who had one episode of wheezing or received bronchodilator therapy for a single episode of illness in the first year of life but who have not had any additional wheezing episodes or bronchodilator therapy for at least 12 months may be enrolled.
* Member of a household that contains an immunocompromised individual
* Member of a household that contains infants less than 6 months of age
* Attends day care with infants less than 6 months of age, and whose parent/guardian is unable or unwilling to suspend daycare for 14 days following immunization. NOTE: Children who attend facilities that separate children by age and minimize opportunities for transmission of virus through direct physical or aerosol contact are acceptable.

Temporary Exclusion Criteria:

The following are temporary or self-limiting conditions. Once resolved, the participant may be enrolled, if otherwise eligible, and if the period of temporary exclusion has been less than 42 days from screening. Otherwise, the participant will need to be rescreened.

* Participant has a rectal temperature of greater than or equal to 100.4°F on the day of planned vaccination, or URI (rhinorrhea, cough, or pharyngitis) or nasal congestion significant enough to interfere with successful vaccination, or otitis media
* Participant has received any killed vaccine or live attenuated rotavirus vaccine within the last 2 weeks, any other live vaccine within the last 4 weeks, or gamma globulin (or other antibody products) within the past 3 months
* Receipt of another investigational vaccine or investigational drug within the prior 28 days of receiving the study inoculation
* Participant has received antibiotics or systemic or nasal steroid therapy for acute illness within the previous 3 days prior to vaccination. NOTE: Permitted concomitant medications include nutritional supplements, medications for gastroesophageal reflux, eye drops, and topical medications, including (but not limited to) topical steroids, topical antibiotics, and topical antifungal agents.
* Participant has received salicylate (aspirin) or salicylate-containing products within the past month
* Participant born at less than 37 weeks gestation and is currently less than 1 year of age

Ages: 6 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3 (Actual)
Dates: Start 2014-09; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Frequency of vaccine-related solicited adverse events (AEs) that occur during the acute monitoring phase of the study, the first 28 days after inoculation | Measured through Day 28
Proportion of participants that develop 4-fold or greater rises in RSV neutralizing antibody titer following vaccination | Measured through Day 56
  Antibody responses to the RSV F glycoprotein will also be assessed by enzyme-linked immunosorbent assay (ELISA).
Severity of vaccine-related solicited AEs that occur during the acute monitoring phase of the study, the first 28 days after inoculation | Measured through Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Ruth A. Karron, MD, Principal Investigator — Center for Immunization Research (CIR), Johns Hopkins Bloomberg School of Public Health (JHSPH)
Locations (1):
- Center for Immunization Research, JHU, Baltimore, Maryland, United States

REFERENCES:
- [Derived] McFarland EJ, Karron RA, Muresan P, Cunningham CK, Valentine ME, Perlowski C, Thumar B, Gnanashanmugam D, Siberry GK, Schappell E, Barr E, Rexroad V, Yogev R, Spector SA, Aziz M, Patel N, Cielo M, Luongo C, Collins PL, Buchholz UJ; International Maternal Pediatric Adolescent AIDS Clinical Trials (IMPAACT) 2000 Study Team. Live-Attenuated Respiratory Syncytial Virus Vaccine Candidate With Deletion of RNA Synthesis Regulatory Protein M2-2 is Highly Immunogenic in Children. J Infect Dis. 2018 Apr 11;217(9):1347-1355. doi: 10.1093/infdis/jiy040. PMID 29509911